CLINICAL TRIAL: NCT07043777
Title: A Retrospective Chart-Review Evaluating Bilateral Modified Catheter Antegrade Cerebral Perfusion Versus Conventional Perfusion in Type A Aortic Dissection Surgery at CMUH (2021-2025)
Brief Title: Effectiveness of Bilateral Modified Catheter Antegrade Cerebral Perfusion in Acute Type A Aortic Dissection Surgery
Acronym: Modified bACP
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH114-REC1-089
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Acute Type A Aortic Dissection
Keywords: Bilateral Modified Catheter Antegrade Cerebral Perfusion; Modified bACP; Cerebral Protection; Neurologic Complications; Retrospective Cohort; Cardiovascular Surgery; China Medical University Hospital; Ascending Aortic Graft Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modified bACP Group: Patients who underwent acute type A aortic dissection repair between 1 Jan 2021 and 30 Apr 2025 using the bilateral modified catheter antegrade cerebral perfusion (Modified bACP) technique.
  Interventions: Procedure: Modified Catheter Antegrade Cerebral Perfusion (Modified bACP)
- Conventional Perfusion Group: Patients who underwent acute type A aortic dissection repair in the same period using the conventional cerebral perfusion strategy (e.g., standard bilateral ACP or surgeon-preferred method). Serves as the comparison cohort.
  Interventions: Procedure: Conventional Brain Perfusion

INTERVENTIONS:
Procedure: Modified Catheter Antegrade Cerebral Perfusion (Modified bACP) — Bilateral modified catheter antegrade cerebral perfusion technique applied during acute type A aortic dissection repair; avoids additional right-axillary incision while providing continuous cerebral flow.
  Groups: Modified bACP Group
Procedure: Conventional Brain Perfusion — Conventional cerebral perfusion strategy (e.g., standard bilateral antegrade cerebral perfusion) used during arch repair according to surgeon preference.
  Groups: Conventional Perfusion Group

SUMMARY:
This single-center retrospective cohort study examines whether a Bilateral Modified Catheter Antegrade Cerebral Perfusion (Modified bACP) technique improves early clinical outcomes in adults undergoing emergency repair of acute Type A aortic dissection (ATAAD).

Electronic medical records at China Medical University Hospital (CMUH) will be reviewed for all ATAAD operations performed between 1 January 2021 and 30 April 2025. Patients treated with Modified bACP will be compared with those managed by conventional perfusion strategies.

The primary outcome is in-hospital stroke. Secondary outcomes include postoperative neurologic deficit, in-hospital mortality, 30-day mortality, hospital and ICU length of stay, mechanical-ventilation duration, need for tracheostomy, acute kidney injury, dialysis requirement, reoperation for bleeding, sepsis, atrial fibrillation, and myocardial infarction.

Findings will clarify the efficacy and safety of Modified bACP and may inform future cerebral-protection protocols in aortic surgery.

DETAILED DESCRIPTION:
Background and Rationale Acute Type A aortic dissection (ATAAD) is life-threatening and requires immediate surgical repair. During hypothermic circulatory arrest, neurologic injury remains a major concern. Conventional bilateral antegrade cerebral perfusion (bACP) provides brain protection but often requires an additional right-axillary arterial cannulation. Our center developed a Modified bACP technique that employs balloon-tipped catheters introduced directly into both carotid arteries, avoiding the extra axillary incision while aiming to maintain stable cerebral flow.

Objectives Primary - To determine whether Modified bACP reduces the incidence of in-hospital stroke compared with conventional perfusion.

Secondary - To evaluate the effect of Modified bACP on early mortality and major postoperative morbidities, and to quantify ICU / hospital resource utilization.

Study Design Design: Retrospective chart review; observational cohort. Setting: China Medical University Hospital, Taichung, Taiwan. Population: All consecutive adult (≥ 18 y) patients who underwent ATAAD repair between 2021-01-01 and 2025-04-30.

Groups:

Modified bACP Group - bilateral modified catheter antegrade cerebral perfusion. Conventional Perfusion Group - standard bilateral ACP or surgeon-selected alternative.

Data Collection Demographics, comorbidities, operative details (CPB time, circulatory-arrest temperature / duration), and postoperative outcomes will be extracted from the electronic medical record by a trained research team and de-identified before analysis.

Outcome Measures Primary - In-hospital stroke (clinical deficit or imaging-confirmed cerebrovascular accident).

Secondary -

* Postoperative neurologic deficit
* In-hospital mortality
* 30-day all-cause mortality
* Hospital length of stay (days)
* ICU length of stay (days)
* Mechanical-ventilation duration (hours)
* Need for tracheostomy
* Acute kidney injury (KDIGO criteria)
* Dialysis requirement
* Reoperation for bleeding
* Sepsis (Sepsis-3)
* Atrial fibrillation (new-onset)
* Myocardial infarction (biomarker + ECG / clinical)

Statistical Analysis Baseline differences will be balanced using inverse-probability weighting of the propensity score derived from age, sex, comorbidities, and operative variables. Logistic or linear regression models will estimate adjusted effect sizes (odds ratios or mean differences) with 95 % confidence intervals. Sensitivity analyses will test robustness to residual confounding. A two-sided P < 0.05 will be considered statistically significant.

Ethics and Oversight The protocol (MACP-2024-03; CMUH114-REC1-089) was approved by the CMUH Research Ethics Committee on 23 May 2025. All data are retrospectively collected and anonymized; informed consent was waived. No U.S. FDA-regulated product or IND/IDE is involved. Because this is a chart review, a formal data-monitoring committee is not required.

Significance By analyzing an extended 2021-2025 cohort, the study increases statistical power to detect clinically relevant differences. Results may validate Modified bACP as a less invasive yet effective cerebral-protection strategy, guiding surgical practice and future prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) who underwent acute Type A aortic dissection repair at China Medical University Hospital between 01 Jan 2021 and 30 Apr 2025.

Exclusion Criteria:

* Documented preoperative stroke or severe neurological deficit prior to surgery.
* Pregnant patients.
* Patients < 18 years old.
* Insufficient or missing medical records that preclude data analysis or verification of outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients treated for acute Stanford Type A aortic dissection with open surgical repair at a single tertiary medical center (China Medical University Hospital, Taichung, Taiwan) between 2021-01-01 and 2025-04-30. The population comprises two retrospectively identified cohorts based on intra-operative cerebral-perfusion strategy (modified bilateral catheter ACP vs conventional perfusion).
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Stroke | Through hospital discharge (average about 14 days post-surgery)
  New-onset cerebrovascular accident or imaging-confirmed stroke occurring after surgery and before hospital discharge. Diagnosis based on neurological examination and/or postoperative brain CT/MRI.

SECONDARY OUTCOMES:
Postoperative Neurological Deficit | Through hospital discharge (average about 14 days post-surgery)
  Any persistent neurological deficit (e.g., motor or sensory loss) documented after surgery and before hospital discharge.
30-Day Mortality | Assessed at 30 days post-surgery
  All-cause mortality occurring within 30 days after the surgical procedure.
Hospital Length of Stay | From end of surgery to discharge (max 30 days)
  Total number of days from operation date to date of hospital discharge.
ICU Length of Stay | From end of surgery to ICU discharge (max 14 days)
  Number of days from ICU admission after surgery until ICU discharge.
Mechanical Ventilation Duration | From end of surgery until extubation (max 120 hours)
  Total hours of invasive mechanical ventilation post-operatively.
Postoperative Acute Kidney Injury (AKI) | Through index hospitalization (average 10-14 days)
  AKI defined by KDIGO criteria based on serum creatinine or urine output during hospitalization. KDIGO stages 0-3 (0 = no injury; 3 = worst). Higher stage = worse renal function.
Dialysis Requirement | Through index hospitalization (average 10-14 days)
  Proportion of patients requiring renal replacement therapy post-operatively.
Number of Participants Requiring Re-operation for Bleeding | Through index hospitalization (average 72 hours)
  Patients requiring return to OR for bleeding or hematoma evacuation.
Number of Participants with Sepsis (Sepsis-3) | Through index hospitalization (average within 7 days)
  Sepsis per Sepsis-3 definition (infection + organ dysfunction) during hospital stay.
Number of Participants with Postoperative Atrial Fibrillation | Through index hospitalization (average within 7 days)
  New-onset atrial fibrillation or arrhythmia episodes requiring treatment.
Myocardial Infarction | Through index hospitalization (average 10-14 days)
  Post-operative MI confirmed by ECG changes and cardiac biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: En-Bo Wu, M.D., Principal Investigator — Department of Anesthesiology, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because institutional privacy policies and the CMUH IRB approval restrict release of de-identified datasets to internal use; any external sharing would require a separate ethics application.

REFERENCES:
- [Background] Pitts L, Kofler M, Montagner M, Heck R, Iske J, Buz S, Kurz SD, Starck C, Falk V, Kempfert J. Cerebral Protection Strategies and Stroke in Surgery for Acute Type A Aortic Dissection. J Clin Med. 2023 Mar 15;12(6):2271. doi: 10.3390/jcm12062271. PMID 36983272